CLINICAL TRIAL: NCT00717795
Title: Physical Activity Intervention for Lung Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fox Chase Cancer Center (Other); University of Alberta (Other); Brown University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-067
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer; Survivor
Keywords: Survivor; Physical Activity; NED; 08-067
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Interviews as Topic; Exercise; Waiting Lists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Arm 1 - Physical Activity intervention
  Interventions: Behavioral: interview and physical activity
- 2: Arm 2 - Wait-list control
  Interventions: Behavioral: interview and wait list

INTERVENTIONS:
Behavioral: interview and physical activity — For Arm 1 participants in the Physical Activity intervention condition will be assessed at baseline, and postintervention Follow-up (at 12 weeks post baseline).
  Groups: 1
Behavioral: interview and wait list — Participants in the control condition (Arm 2)will be assessed at baseline and 12 weeks post baseline (Follow-up). At this time, the PA intervention will be offered at no cost to the participants in the control condition. If the waitlist participant chooses to complete the PA intervention after the 12 week waitlist period, program satisfaction will be assessed after study completion.
  Groups: 2

SUMMARY:
The purpose of this study is to learn how many lung cancer survivors will agree to a physical activity program. We also want to know if lung cancer survivors benefit from this program. This information will help us to develop our services for lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis and treatment at MSKCC of primary NSCLC; and/or pulmonary carcinoid;
* At least one year post thoracic surgical resection;
* Have no evidence of NSCLC or any other cancer at the time of study enrollment and not receiving any cancer treatment;
* Currently sedentary or insufficiently active, defined by the American College of Sports Medicine (ACSM) and the Centers for Disease Control and Prevention as less than a total of 150 minutes of at least moderate intensity PA per week;
* Able to complete a six-minute walk test (6MWT);
* Able to provide informed consent.

FOCUS GROUP ONLY:

• Completed the Physical Activity program offered through this study (08067);

Exclusion Criteria:

* Presence of one of the following medical factors at screening:

  * regular use of an ambulatory aid (cane or walker);
  * resting oxygen saturation less than 88%;
  * inability to walk due to severe arthritis or other musculoskeletal problems;
  * a diagnosis of unstable angina in the previous 6 weeks;
  * a heart attack, angioplasty or heart surgery in the previous 3 months;
  * current heart rate <50 or >120 at rest; current uncontrolled hypertension;
  * current significant valvular heart disease or decompensated congestive heart failure and
  * patient reported pain of any origin that would preclude participation in the proposed PA intervention
* Evidence of significant medical cognitive or psychiatric disturbance sufficient, in the investigator's judgment, to preclude participation in the intervention
* Self-reporting of greater than 60 minutes of vigorous activity per week or 150 minutes of moderate intensity PA per week.
* Patient resides at more than two hours travel distance from the Center
* Insufficient English fluency to complete evaluation tools.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total, we will recruit and enroll a random sample of 70 lung cancer survivors who are at least one year post thoracic surgical resection and have no evidence of NSCLC or any other cancer at the time of study enrollment and not receiving any adjuvant treatment.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-06-10 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility (acceptability, adherence, treatment integrity, retention, participant satisfaction) of implementing a physical activity intervention trial among sedentary and insufficiently active lung cancer survivors. | conclusion of the study

SECONDARY OUTCOMES:
Obtain preliminary data on effect of a physical activity intervention on functional ability, health-related QOL, dyspnea, fatigue, balance, strength & self-report physical activity among sedentary and insufficiently active lung cancer survivors | conclusion of the study
To obtain preliminary data on factors associated with feasibility using variables from Social Cognitive Theory and assess their relationship with treatment adherence and dropout. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org